CLINICAL TRIAL: NCT00402740
Title: Protected Carotid Artery Stenting in Subjects at High Risk for Carotid Endarterectomy (CEA)
Brief Title: Protected Carotid Artery Stenting in Subjects at High Risk for Carotid Endarterectomy (CEA) (PROTECT)
Acronym: PROTECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 640-0071
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Results first posted 2012-06-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-05

CONDITIONS: Carotid Artery Disease
Keywords: Carotid; Artery; Disease; Stent; PROTECT; XACT; EMBOSHIELD
MeSH Terms: conditions — Carotid Artery Diseases; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Xact Stent with either Emboshield Pro (Gen 5) or Emboshield (Gen 3) — All subjects will receive the Xact™ Rapid Exchange Carotid Stent System. The first 220 consecutively enrolled subjects will be treated with the investigational filter system, the Emboshield® Pro Rapid Exchange Embolic Protection System (Generation 5). The remaining subjects will be treated with the FDA approved Emboshield® BareWire™ Rapid Exchange Embolic Protection System (Generation 3).
  Other Names: Xact stent; Emboshield Pro (Gen 5); Emboshield (Gen 3)

SUMMARY:
The purpose of this study is to evaluate the long-term safety and efficacy of the Xact™ Rapid Exchange Carotid Stent System used in conjunction with the Emboshield® Pro Rapid Exchange Embolic Protection System (Generation 5) and the Emboshield® BareWire™ Rapid Exchange Embolic Protection System (Generation 3), in the treatment of atherosclerotic carotid artery disease in high-surgical risk subjects.

ELIGIBILITY:
Inclusion Criteria Subject must be ≥ 18 years of age.

Subject has the ability to cooperate with study procedures and agrees to return for all required follow-up visits, tests and exams.

Female subjects of childbearing potential must have a documented negative pregnancy test within 30 days prior to the index procedure.

Subjects taking warfarin may be included if their dosage is reduced before the index procedure to result in an INR of 1.5 or less. Warfarin may be restarted to therapeutic dose after the index procedure.

The subject must sign a written informed consent prior to the initiation of any study procedures, using a form that is approved by the Institutional Review Board (IRB) or Medical Ethics Committee (EC).

The life expectancy of the subject is at least two years.

The subject has a lesion located in the internal carotid artery (ICA); the carotid bifurcation may be involved.

The target lesion is intended to be treated with a single stent.

Target ICA vessel diameter must be visually estimated to be:

* ≥2.5 mm and ≤7.0 for the Emboshield Pro (Gen 5)
* ≥ 2.8 mm and ≤6.2 for the Emboshield (Gen 3)

And

* ≥4.0 mm and ≤9.0 mm for the Xact Stent treatment area.

The subject has a carotid artery stenosis determined by ultrasound or angiography (visual estimate) to be:

* ≥50% for symptomatic subjects

Or

* ≥80% for asymptomatic subjects

High-risk inclusion criteria for either anatomical or co-morbid risk factors are present. The subject must fulfill at least one of the criteria, Category I or II risk factors, listed below to meet the inclusion criteria.

Category I Anatomic Risk Factors

* Previous radiation treatment to the neck or radical neck dissection
* Target lesion is at or above the second vertebral body C2 (level of jaw)
* Inability to extend the head due to cervical arthritis or other cervical disorders
* Tracheostomy or tracheal stoma
* Laryngectomy
* Contralateral laryngeal nerve palsy
* Severe tandem lesions

Category II Co-morbid Risk Factors

* Previous CEA with significant restenosis (as defined for symptomatic or asymptomatic subjects)
* Total occlusion of the contralateral carotid artery
* Left ventricular ejection fraction < 35%
* Congestive Heart failure New York Heart Association (NYHA) Functional Class III or higher
* Dialysis dependent renal failure
* Canadian Cardiovascular Society Angina Classification III or higher or unstable angina
* Requires coronary artery bypass surgery, cardiac valve surgery, peripheral vascular surgery, or abdominal aortic aneurysm repair within 60 days

  •≥80 years of age
* Myocardial infarction within previous 6 weeks
* Abnormal stress test. Treadmill, thallium or dobutamine echo are acceptable. The stress tests should be sufficiently abnormal to place the subject at increased risk for CEA. This includes subjects with two or more proximal diseased coronary arteries of >70% stenosis that have not or cannot be revascularized or <30 days since revascularization.
* Severe pulmonary disease, including at least one of the following: requires chronic O2 therapy; resting PO2 ≤60 mm Hg, Hematocrit ≥50%, FEV₁ or DLCO ≤50% of normal.

Exclusion Criteria

* The subject is participating in another investigational trial that would interfere with the conduct or result of this study.
* The subject has dementia or a neurological illness that may confound the neurological evaluation.
* Total occlusion of the target vessel.
* There is an existing, previously placed stent in the target artery.
* The subject has a known life-threatening allergy to the contrast media that cannot be treated.
* Subject has history of intolerance or allergic reaction to any of the study medications including aspirin, Clopidogrel bisulfate (Plavix®) or Ticlopidine (Ticlid®), heparin or Bivalirudin (Angiomax™). Subjects must be able to tolerate a combination of aspirin and Clopidogrel or aspirin and Ticlopidine.
* The subject has a GI bleed that would interfere with antiplatelet therapy.
* The subject has known cardiac sources of emboli, including but not limited to current or past history of paroxysmal or sustained atrial fibrillation (treated or untreated), valve replacement, etc.
* Subject has Hemoglobin (Hgb) less than 8 gm/dL (unless on dialysis), platelet count <50,000/mm3, or known heparin associated thrombocytopenia.
* The subject has a history of bleeding diathesis or coagulopathy including thrombocytopenia or an inability to receive heparin or Bivalirudin (Angiomax™) in amounts sufficient to maintain an ACT of >250, or will refuse blood transfusion.
* The subject has atherosclerotic disease involving adjoining vessels that precludes safe placement of the guiding catheter or sheath.
* The subject has other abnormal angiographic findings that indicate the subject is at risk for a stroke due to a problem other than that of the target lesion, such as: ipsilateral arterial stenosis greater in severity than the target lesion, cerebral aneurysm, or arteriovenous malformation of the cerebral vasculature.
* There is evidence of a carotid artery dissection prior to the initiation of the index procedure.
* There is an angiographically visible thrombus.
* There is any condition that precludes proper angiographic assessment, placement of the cerebral protective system or makes percutaneous arterial access unsafe, e.g. morbid obesity, sustained systolic blood pressure >180 mm Hg, tortuosity, occlusive disease, vessel anatomy, or aortic arch anatomy.
* Occlusion (TIMI 0 flow), or string sign of the ipsilateral common or internal carotid artery.
* There is evidence of bilateral carotid stenosis that would require intervention within 30 days of the index procedure.
* There is evidence of a stroke within the previous 30 days of the index procedure.
* There is a planned treatment of a non-target lesion within 30 days post-index procedure.
* There is a history of intracranial hemorrhage within the previous 3 months, including hemorrhagic transformation of an ischemic stroke.
* There is a history of an ipsilateral stroke with fluctuating neurologic symptoms within one year of the index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2006-11; Primary Completion 2011-06 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seemant Chaturvedi, MD, Study Chair — Wayne State University Stroke Program; William A Gray, MD, Study Chair — Columbia University; Jon Matsumura, MD, Study Chair — University of Wisconsin, Madison
Locations (38):
- United States (38):
  - Washington Hospital, Fremont, California
  - El Camino Hospital, Mountain View, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Stanford University Medical Center, Stanford, California
  - University of Connecticut Health Center, Farmington, Connecticut
  - Memorial Hospital Jacksonville, Jacksonville, Florida
  - Lakeland Regional Medical Center, Lakeland, Florida
  - Munroe Regional Medical Center, Ocala, Florida
  - Hawaii Permanente Medical Group-Kaiser Foundation Hospital, Honolulu, Hawaii
  - Northwestern University Memorial Hospital, Chicago, Illinois
  - St. John's Hospital / Memorial Medical Center, Springfield, Illinois
  - Parkview Hospital, Fort Wayne, Indiana
  - St. Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - McLaren Regional Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Our Lady of Lourdes Medical Center, Camden, New Jersey
  - St. Michael's Medical Center, Newark, New Jersey
  - Millard Fillmore Hospital-Kaleida Health Systems, Buffalo, New York
  - Lenox Hill Hospital, New York, New York
  - WakeMed Hospital, Raleigh, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Pinnacle Health Hospital, Harrisburg, Pennsylvania
  - St. Joseph's Medical center, Wyomissing, Pennsylvania
  - Greenville Memorial Medical Center, Greenville, South Carolina
  - Holston Valley Medical Center, Kingsport, Tennessee
  - Mercy Medical Center West / Baptist Hospital of East Tennessee, Knoxville, Tennessee
  - Austin Heart P.A., Austin, Texas
  - Presbyterian Heart Institute, Dallas, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - Chesapeake General Hospital, Norfolk, Virginia
  - Bon Secours St. Mary's Hospital, Richmond, Virginia
  - St. Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- See also: Results of carotid artery stenting with distal embolic protection with improved systems: Protected Carotid Artery Stenting in Patients at High Risk for Carotid Endarterectomy (PROTECT) trial. — http://www.ncbi.nlm.nih.gov/pubmed/22236885

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 322 subjects were enrolled in the PROTECT study at 38 clinical sites in the United States. The first subject was enrolled on November 29, 2006, and enrollment was completed on June 18, 2008.
Period: Overall Study
Arm/Group | Group 1
Started | 322
Completed | 242
Not Completed | 80
Not completed — Withdrawal by Subject | 18
Not completed — Death | 50
Not completed — Lost to Follow-up | 6
Not completed — No stent. Completed FU at 30 days. | 5
Not completed — Subject disposition unknown. | 1

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 322
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 71
  >=65 years | 251
Age Continuous [Mean (Standard Deviation); unit: years] | 72.7 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115
  Male | 207
Region of Enrollment [Number; unit: participants]
  United States | 322

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimate of Freedom From the Composite of Any Death, Stroke and MI During the 30 Day Post Procedural Period (DSMI), Plus Fatal and Non-fatal Ipsilateral Stroke From 31-365 Days and Annually Thereafter for a Total of 3 Years.
Description: Freedom from DSMI to 30 days or ipsilateral stroke from 31 days to 3 years. KM event free (%) curve.
Time Frame: 3 years
Population: Intent to Treat (ITT)
Measure: Number; unit: Event-free percentage
Groups:
- Group 1: Includes only the most serious event for each subject and includes only each subject's first occurrence of the event.
Arm/Group | Group 1
Number analyzed (Participants) | 322
Event-free percentage | 95.5 [1.72 to 6.03]

2. Secondary Outcome: Acute Device Success
Description: Defined by the attainment of <50% residual stenosis covering an area no longer than the original lesion treated with the stent.
Time Frame: Post-procedure
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Xact Stent: The Xact stent success were counted per subject
- Emboshield Pro Gen 5: Participants receiving Emboshield Pro Gen 5. Emboshield Pro success were counted per filter.
- Emboshield Gen 3: Participants receiving Emboshield Gen 3 Emboshield Gen3 success were counted per filter.
Arm/Group | Xact Stent | Emboshield Pro Gen 5 | Emboshield Gen 3
Number analyzed (Participants) | 317 | 222 | 101
percentage of participants | 98.7 [96.80 to 99.66] | 97.3 [94.21 to 99.00] | 97.0 [91.56 to 99.38]

3. Secondary Outcome: Procedural Success
Description: Defined as the attainment of less than 50% residual stenosis (per angiographic core lab) of the target lesion and the absence of DSMI at 30 days post-index procedure.
Time Frame: 30 Days
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1
Number analyzed (Participants) | 322
percentage of participants | 95.30 [92.43 to 97.37]

4. Secondary Outcome: Composite of Any Transient Ischemic Attack (TIA) and Amaurosis Fugax
Description: Includes only each subject's first occurrence of each event.
Time Frame: ≤30 days
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1
Number analyzed (Participants) | 322
percentage of participants | 2.8 [1.29 to 5.24]

5. Secondary Outcome: Kapan-Meier Estimate of Freedom From Clinically Driven Target Lesion Revascularization Through Three Years.
Time Frame: 3 years
Population: ITT
Measure: Number; unit: Event-free percentage
Arm/Group | Group 1
Number analyzed (Participants) | 317
Event-free percentage | 98.2

ADVERSE EVENTS:
Time Frame: Three years post-procedure
Description: Organ systems designations were chosen to match Abbott Categories coding as closely as possible and may differ from other coding systems.
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 221/313
Other Adverse Events (participants affected / at risk) | 236/313
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=313)
Hematoma (Injury, poisoning and procedural complications) | 2 (2) — Access site complication
Occlusion (Injury, poisoning and procedural complications) | 2 (2) — Access site complication
Epistaxis (Surgical and medical procedures) | 5 (5) — Bleeding
Gastrointestinal (Gastrointestinal disorders) | 14 (15) — Bleeding
Hematuria (Surgical and medical procedures) | 3 (3) — Bleeding
Oropharyngeal (Surgical and medical procedures) | 1 (1) — Bleeding
Other (Injury, poisoning and procedural complications) | 3 (3) — Bleeding
Anemia (Blood and lymphatic system disorders) | 27 (27) — Blood dyscrasia
Leukopenia (Blood and lymphatic system disorders) | 1 (1) — Blood dyscrasia
Abnormal lab test (Cardiac disorders) | 1 (1) — Cardiac
Angina (Cardiac disorders) | 10 (15) — Cardiac
Arrhythmia (Cardiac disorders) | 30 (46) — Cardiac
Cardiac arrest (Cardiac disorders) | 11 (11) — Cardiac
Congestive heart failure (Cardiac disorders) | 30 (41) — Cardiac
Coronary artery diseasee (Cardiac disorders) | 39 (51) — Cardiac
Hypertensive cardiovascular disease (Cardiac disorders) | 1 (1) — Cardiac
Myocardial infarctionsee (Cardiac disorders) | 13 (13) — Cardiac
Structural heart disease (Cardiac disorders) | 14 (15) — Cardiac
Hypertension (Renal and urinary disorders) | 9 (9) — Hemodynamic
Hypotension (Cardiac disorders) | 6 (6) — Hemodynamic
Presyncope /syncope (General disorders) | 3 (3) — Hemodynamic
Syncope (General disorders) | 6 (8) — Hemodynamic
Myocardial infarction Non Q wave (Cardiac disorders) | 2 (2) — Myocardial infarction
Amaurosis fugax (Nervous system disorders) | 1 (1) — Neurologic other than stroke
Confusion (Nervous system disorders) | 2 (2) — Neurologic other than stroke
Hyperperfusion syndrome (Nervous system disorders) | 1 (1) — Neurologic other than stroke
Neurologic other (Nervous system disorders) | 21 (26) — Neurologic other than stroke ??I'll require a little more information.
Seizure (Nervous system disorders) | 3 (4) — Neurologic other than stroke
Subdural hematoma (Skin and subcutaneous tissue disorders) | 1 (1) — Neurologic other than stroke
Transient Ischemic Attack (Nervous system disorders) | 11 (12)
Visual disturbance (Nervous system disorders) | 2 (4) — ?? or eye disorders ??
Anemia (Blood and lymphatic system disorders) | 8 (8)
Arrhythmia (Cardiac disorders) | 8 (8) — ?Procedure related? or neurological?
Cardiac arrest (Cardiac disorders) | 1 (1) — Procedure related
Dissection (Injury, poisoning and procedural complications) | 1 (1) — Procedure related
Fluid overload (Injury, poisoning and procedural complications) | 1 (1) — Procedure related
Hypertension (Injury, poisoning and procedural complications) | 1 (1) — Procedural
Hypotension (Injury, poisoning and procedural complications) | 26 (26) — Procedure related
Pain (Injury, poisoning and procedural complications) | 1 (1) — Procedure related?
Urinary retention (General disorders) | 1 (1) — ?Procedure related?
Ipsilateral major (Nervous system disorders) | 3 (3) — Stroke
Ipsilateral minor (Nervous system disorders) | 8 (8) — Stroke
Aneurysm (Vascular disorders) | 3 (3) — Vascular
Deep vein thrombosis (Vascular disorders) | 4 (4) — Vascular
Dissection (Injury, poisoning and procedural complications) | 1 (2) — Vascular
Instent restenosis (Injury, poisoning and procedural complications) | 7 (9) — Vascular
Peripheral vascular disease (Vascular disorders) | 23 (30) — Vascular
Pseudoaneurysm (Vascular disorders) | 1 (1) — Vascular
Restenosis (Vascular disorders) | 1 (1) — Vascular
Stenosis (Vascular disorders) | 11 (12) — Vascular
Thrombosis (Vascular disorders) | 2 (2) — Vascular
Allergic reaction (General disorders) | 1 (1) — Other
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 26 (32) — Other
Gastrointestinal (Gastrointestinal disorders) | 32 (50) — Other
Genitourinarynal (Renal and urinary disorders) | 26 (34) — Other
Infection (Infections and infestations) | 26 (33) — Other
Mental health related (Psychiatric disorders) | 1 (1) — Other
Metabolic (Metabolism and nutrition disorders) | 14 (18) — Other
Miscellaneous (General disorders) | 5 (5) — Other
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 29 (33) — Other
Respiratory (Respiratory, thoracic and mediastinal disorders) | 55 (91) — Other
Trauma (Psychiatric disorders) | 5 (6) — Other
Non-ipsilateral major (Vascular disorders) | 5 (5) — Stroke
Non-ipsilateral minor (Vascular disorders) | 4 (5) — Stroke
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=313)
Anemia (Blood and lymphatic system disorders) | 20 (23)
Arrhythmia (Cardiac disorders) | 25 (27)
Neurologic other (Nervous system disorders) | 37 (51) — ??Neurologic other than stroke?? I may need additional description
Arrhythmia (Cardiac disorders) | 22 (24) — Procedure related
Headache (General disorders) | 17 (18) — Procedure related
Hypotension (Cardiac disorders) | 43 (45) — Procedure related
Nausea/vomiting (General disorders) | 17 (17) — Procedure related
Pain (Injury, poisoning and procedural complications) | 30 (36) — Procedure related
Peripheral vascular disease (Vascular disorders) | 28 (34) — Procedure related
Other: Gastrointestinal (Gastrointestinal disorders) | 48 (98)
Other: Genitourinary (General disorders) | 43 (63)
Other: Infection (Infections and infestations) | 31 (52)
Other: Metabolic (General disorders) | 28 (36)
Other: Miscellaneous (General disorders) | 63 (118) — ?? i'll need additional description
Other: Musculoskeletal (Musculoskeletal and connective tissue disorders) | 67 (122)
Other: Respiratory (Respiratory, thoracic and mediastinal disorders) | 55 (80)
Other: Trauma (General disorders) | 16 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator (PI), Institute, and Research Site (RS) acknowledge this is a multi-center study. An independent, joint publication is anticipated from investigators in the study, including the PI. Therefore, the PI, Institute, and RS agree not to publish or present the results before the publication of the multi-center investigator paper, but in no event shall PI, Institute, and/or RS be so restricted after the expiration of twelve months from completion of the Study at all sites.